CLINICAL TRIAL: NCT00216645
Title: Open-label Study to Verify Effectiveness, Safety of Pegylated Liposomal Doxorubicin 50 mg/m2 Administered Every 4 Weeks to Patients With Mullerian Carcinoma (Epithelial Ovarian Carcinoma, Primary Carcinoma of Fallopian Tube, Peritoneal Carcinoma) Who Have Undergone Prior Platinum-based Chemotherapy.
Brief Title: Phase II Clinical Study of Pegylated Liposomal Doxorubicin Hydrochloride Injection as 2nd-line or Later Therapy in Patients With Mullerian Carcinoma (Epithelial Ovarian Carcinoma, Primary Carcinoma of Fallopian Tube, Peritoneal Carcinoma) Having Prior Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004867
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Ovarian Neoplasms
Keywords: Müllerian Carcinoma; Doxil; Japanese Patients
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Doxorubicin

INTERVENTIONS:
Drug: doxorubicin hydrochloride

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of pegylated liposomal doxorubicin hydrochloride injection in Japanese patients with Mullerian carcinoma. This clinical study is a multi-center, non-randomized, open-label study in Japanese patients with Mullerian carcinoma (including epithelial ovarian carcinoma, primary carcinoma of fallopian tube, peritoneal carcinoma) with a prior history of platinum-based chemotherapy. Eighty patients will be administered intravenously at least two cycles of 50 mg/m2 of pegylated liposomal doxorubicin hydrochloride every 4 weeks to investigate the effectiveness and safety of the treatment.

DETAILED DESCRIPTION:
Pegylated liposomal Doxorubicin hydrochloride is intended to change the pharmacokinetics of conventional doxorubicin in the blood and to improve the safety and effectiveness of the drug. Pegylated liposomal doxorubicin hydrochloride has been approved in many countries including US and EU, becoming a standard drug for 2nd-line therapy in ovarian cancer and AIDS-related Kaposi's Sarcoma. This clinical study was planned to assess effectiveness and safety for Japanese patients with Müllerian carcinoma (including epithelial ovarian carcinoma, primary carcinoma of fallopian tube, peritoneal carcinoma), who had a prior history of receiving platinum-based chemotherapy such as Cisplatin (which is considered to be the standard chemotherapy for ovarian carcinoma). In this study, at least two cycles of pegylated liposomal doxorubicin hydrochloride 50 mg/m2 will be intravenously administered to 80 patients every 4 weeks. These patients include twenty 2nd-line "platinum-sensitive" and sixty "platinum-resistant" 2nd-line or 3rd-line patients. Pegylated liposomal doxorubicin hydrochloride 50 mg/m2 will be given by intravenous drip infusion on day 1. After this, a 27-day drug-free period will be followed as one cycle. At least two cycles will be given as long as the patient does not meet the discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian cancer who had a response to initial treatment but then relapsed within 12 months are eligible
* Patients with ovarian cancer who have received one or two prior chemotherapy treatment are eligible
* Patients must have measurable disease, good performance status and adequate major organ function

Exclusion Criteria:

* Patients with concomitant disease that may affect the conduct of the study and the evaluation of pegylated liposomal doxorubicin hydrochloride
* Patients with systemic infection
* Patients with active second cancer besides the ovarian cancer
* Patients with pleural effusion or ascites requiring continuous drainage at the time of enrollment
* Patients with pericardial fluid requiring drainage
* Patients with myocardial infarction and/or angina attack within 90 days prior to enrollment.

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate as antitumor effect (tumor shrinkage)

SECONDARY OUTCOMES:
The incidence and the severity of adverse events and adverse drug reactions; the median time to response and median duration of response and these ranges in response patients

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: Phase 2 Clinical study of JNS002 ( DOXILTM ) in patients with Mullerian Carcinoma (epithelial ovarian carcinoma,primary carcinoma of fallopian tube,peritoneal carcinoma ) Having a Therapeutic History of Platinum-Based Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=405&filename=CR004867_CSR.pdf